CLINICAL TRIAL: NCT04005183
Title: Molecular Dissection of the Renal Cell Carcinoma Tumor Microenvironment for the Discovery of Novel Therapeutic Targets
Brief Title: Renal Cell Carcinoma Microenvironment Discovery Project
Acronym: REMEDY
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Celsius Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-5204
Record Dates: First submitted 2019-05-20; First posted 2019-07-02 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Genomics; Single-cell; Microenvironment; Immunotherapy; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Kidney Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Kidney Diseases; Urologic Diseases
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Kidney Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Kidney Diseases; Urologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy, surgically resected tumour specimen, blood, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Patients undergoing nephrectomy at the University Health Network are eligible for enrolment. All renal cell carcinoma histological subtypes and stages are eligible. Tumor, blood and urine samples are acquired at the time of nephrectomy.

SUMMARY:
This study will obtain tumor samples from nephrectomy specimens in a multi-regional fashion and subject them to integrated genomics, proteomics, pathological, and radiological assessment. The goal is to better understand the the molecular basis for how various cells within the tumor microenvironment act in a coordinated manner to facilitate tumor progression and therapy resistance. Our ultimate aim is to leverage this data resource to identify novel therapeutic targets and biomarkers to improve the clinical management of this disease.

DETAILED DESCRIPTION:
This study is an observational prospective trial where renal cell carcinoma samples are isolated from nephrectomy specimens in a multi-regional manner and subjected to an integrated genomic, proteomic, pathological, radiological assessment to provide a detailed morphological and molecular view of the RCC microenvironment.

The major genomics technologies used to examine tumour specimens include single cell RNA sequencing including nuclear (NUCseq) and epitope sequencing (CITEseq). Additionally, bulk RNA/DNA sequencing, targeted mutational profiling, and imaging mass cytometry will be performed. These technologies will determine mutational and gene/protein expression profiles of various heterogeneous cell populations within the tumour microenvironment, including cancer, immune, and supporting cells. This will allow identification of mutations and abnormal expression patterns within individual cells, that will be used to infer targetable vulnerabilities and biomarker signatures.

ELIGIBILITY:
Inclusion Criteria:

* Nephrectomy
* Primary or metastatic disease
* Any histology of renal cell carcinoma

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic Renal cell carcinoma undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Molecular profiling of various cell populations within tumour by using single cell RNAseq. | 10 years
  The RNA transcripts of tumour cells will be sequenced and subjected to informatics and descriptive statistical methods to generate comprehensive data sets that aid in better understanding of the tumour microenvironment in various patients and disease types. These data sets will provide insights into drug target discovery, and used as hypothesis-generating guidance for future study aims.
Determination of the radiological and pathological features associated with the derived tumor microenvironment molecular data | 10 years
  The radiological and pathological assessment on each tumour case will be paired with the gene- and protein-level data to provide a comprehensive picture of the disease. These datasets will be used as training sets to guide machine learning technologies with the intention of aiding diagnosis, prognosis prediction, and treatment plans in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Finelli, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada

DOCUMENTS (2):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT04005183/Prot_000.pdf
  • Informed Consent Form (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT04005183/ICF_001.pdf